CLINICAL TRIAL: NCT01205503
Title: Randomized, Blinded Trial of Mesna to Prevent Doxorubicin-induced Plasma Protein Oxidation and TNF-α Release
Brief Title: Trial of Mesna to Prevent Doxorubicin-induced Plasma Protein Oxidation and Tumor Necrosis Factor Alpha (TNF-α) Release
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mara Chambers (Other)
Responsible Party: Sponsor-Investigator, Mara Chambers, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0431-F1V
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer; Non-Hodgkin's Lymphoma
Keywords: chemobrain; Oxidative Stress; Mesna
MeSH Terms: conditions — Breast Neoplasms; Lymphoma, Non-Hodgkin; Chemotherapy-Related Cognitive Impairment | interventions — Mesna; Sodium Chloride; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycle 1 Saline; Cycle 2 Mesna (Other): Saline infused over 15 minutes administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) with following Cyclophosphamide 6 hours post doxorubicin during 1st cycle, then Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion with following Cyclophosphamide 6 hours post doxorubicin during 2nd cycle
  Interventions: Drug: Mesna; Drug: Saline; Drug: Doxorubicin; Drug: Cyclophosphamide
- Cycle 1 Mesna; Cycle 2 Saline (Other): Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion with following Cyclophosphamide 6 hours post doxorubicin during 1st cycle, then Saline administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) with following Cyclophosphamide 6 hours post doxorubicin during 2nd cycle
  Interventions: Drug: Mesna; Drug: Saline; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Mesna — Mesna: 360 mg/m2 in 50 mL normal saline (NS) either on cycle 2 or cycle 1, day 1. Infused over 15 minutes
  Other Names: Mesnex
Drug: Saline — Saline (used as a placebo) infused over the same time as mesna intervention
  Other Names: Placebo
Drug: Doxorubicin — 60mg/m2 given IV over 15 minutes after receiving mesna or saline. Can allow for premedications of Ondansetron 8 mg orally, dexamethasone 12 mg orally, Aprepitant 125 mg orally.
  Other Names: Adriamycin
Drug: Cyclophosphamide — 600 mg/m2 IV over 30 minutes. Start 6 hours after doxorubicin started.
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cycloblastin

SUMMARY:
The purpose of this study is to determine whether the drug mesna is able to block a series of chemical changes that occur in the blood of patients who receive the chemotherapy medicine doxorubicin. The researchers believe these blood chemical changes may the cause of "cloudy thinking" or "chemobrain" that are reported by some patients receiving chemotherapy.

DETAILED DESCRIPTION:
Patients with lymphoma and breast cancer receiving chemotherapy regimens that include anthracycline drugs, such as doxorubicin, are at risk for developing cognitive and cardiac impairment. This potential cognitive impairment is refered to as "chemobrain" by some patients. We have demonstrated in mice that the drug mesna, which is used to prevent other complications of other chemotherapy drugs, prevents certain types of doxorubicin-induced damage of blood proteins. Blocking doxorubicin's damage of these blood proteins has blunted or prevented the subsequent markers of neurologic and cardiac injury in mice. This clinical trial will determine if mesna prevents doxorubicin-induced damage of blood proteins in cancer patients, and may establish if blood protein injury is the first step in anthracycline-induced cognitive and cardiac dysfunction and if using the drug mesna can blunt or prevent these changes in blood markers of injury for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

Participants must have histologically or cytologically confirmed breast cancer or non-hodgkin lymphoma and independent of protocol eligibility be determined to require one of the chemotherapy regimens listed below

Participants must require as standard-of-care treatment a chemotherapy regimen that includes one of the following combinations:

* doxorubicin 60 mg/m2 and cyclophosphamide 600 mg/m2;
* doxorubicin 50 mg/m2, cyclophosphamide 500 mg/m2, and docetaxel 75 mg/m2;
* doxorubicin 50 mg/m2, cyclophosphamide 750 mg/m2, vincristine 1.4 mg/m2 (capped at 2 mg dose), and prednisone 100 mg +/- rituximab 375 mg/m2

Age >18 years.Because these treatment regimens are rarely used in pediatric oncology, children are excluded from this study but will be eligible for future pediatric phase 2 trials.

Life expectancy of greater than 6 months.

Zubrod performance score 2 or better.

Patients must have normal organ and marrow function as defined below:

* leukocytes >3,000/microliter (mcL) (unless due to cancer in marrow)
* absolute neutrophil count >1,500/mcL (unless due to cancer in marrow)
* platelets >100,000/mcL (unless due to cancer in marrow)
* total bilirubin <1.5 X normal institutional limits
* Aspartate aminotransferase (AST) or serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase (SGPT) <2.5 X institutional upper limit of normal
* creatinine within normal institutional limits OR
* creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* left ventricular function ≥ 50 % ejection fraction

Because the standard of care chemotherapy agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.

Patients may not be receiving any other investigational agents

Patients with known brain metastases should be excluded from this clinical trial because progressive neurologic dysfunction would confound the evaluation of neuro-cognitive outcomes.

History of allergic reactions attributed to compounds of similar chemical or biologic composition to mesna or other agents used in the study (ie. sulfur containing drugs including "sulfa antibiotics" and celecoxib).

Patients requiring ongoing pharmacologic treatment of dementia are excluded.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Pregnant women are excluded from this study because the chemotherapy agents have known teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued if the mother is treated with chemotherapy.

HIV-positivity is NOT a specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Chambers, M.D., Principal Investigator — Markey Cancer Center
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data is already available as part of the published article supplement. PubMed Identification (ID) # 25909710

REFERENCES:
- [Result] Hayslip J, Dressler EV, Weiss H, Taylor TJ, Chambers M, Noel T, Miriyala S, Keeney JT, Ren X, Sultana R, Vore M, Butterfield DA, St Clair D, Moscow JA. Plasma TNF-alpha and Soluble TNF Receptor Levels after Doxorubicin with or without Co-Administration of Mesna-A Randomized, Cross-Over Clinical Study. PLoS One. 2015 Apr 24;10(4):e0124988. doi: 10.1371/journal.pone.0124988. eCollection 2015. PMID 25909710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at the University of Kentucky Markey Cancer Center in Lexington, Kentucky, USA between October 2010 and May 2012.
Groups:
- Cycle 1 Saline; Cycle 2 Mesna: Saline infused over 15 minutes administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) during 1st cycle, then Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion during 2nd cycle
  Mesna: Mesna: 360 mg/m2 in 50 mL normal saline (NS) on cycle 2, day 1. Infused over 15 minutes
- Cycle 1 Mesna; Cycle 2 Saline: Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion during 1st cycle, then Saline administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) during 2nd cycle
  Mesna: Mesna: 360 mg/m2 in 50 mL normal saline (NS) on cycle 1, day 1. Infused over 15 minutes
Period: First Intervention (1st Cycle)
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Second Intervention (2nd Cycle)
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.81 (11.70) | 51.75 (15.51) | 54.78 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Treatment Type [Number; unit: participants]
  Doxorubicin and cyclophosphamide (AC) | 6 | 5 | 11
  AC, vincristine, and prednisone (CHOP) | 9 | 10 | 19
  Doxorubicin, cyclophosphamide and docetaxel (TAC) | 1 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants]
  0- Fully Active | 10 | 8 | 18
  1- Restricted | 6 | 8 | 14
Cancer Diagnosis [Number; unit: participants]
  Breast | 7 | 6 | 13
  Lymphoma | 9 | 10 | 19
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 2.01 (0.23) | 1.93 (0.26) | 1.97 (0.25)
log TNF Alpha [Mean (Standard Deviation); unit: log(pg/ml)] | 1.27 (1.11) | 1.30 (1.16) | 1.28 (1.12)
log TNF receptor 1 [Mean (Standard Deviation); unit: log(pg/ml)] | 7.29 (0.44) | 7.04 (0.46) | 7.17 (0.46)
Log interleukin (IL)-18 [Mean (Standard Deviation); unit: log(pg/ml)] | 6.06 (0.93) | 6.16 (0.76) | 6.11 (0.84)
Log Protein Carbonyl (PC) [Mean (Standard Deviation); unit: log(nmol/mg protein)] | 4.39 (0.34) | 4.33 (0.38) | 4.36 (0.36)
Log Plasma 4-hydroxynonenal (HNE) [Mean (Standard Deviation); unit: log(pmol/mg)] — This baseline measurement is standardized to the control on the plate and then log transformed. The resulting ratio of plate assay value relative to control can be < 1 resulting in a negative log value.
  log(pmol/mg) | -0.31 (0.22) | -0.28 (0.20) | -0.29 (0.21)
Log 3-nitrotyrosine (3NT) [Mean (Standard Deviation); unit: log(ng/mg protein)] — This baseline measurement is standardized to the control on the plate and then log transformed. The resulting ratio of plate assay value relative to control can be < 1 resulting in a negative log value.
  log(ng/mg protein) | -0.11 (0.26) | -0.05 (0.16) | -0.08 (0.21)
Log TNF Receptor 2 [Mean (Standard Deviation); unit: log(pg/ml)] | 8.31 (0.68) | 8.15 (0.74) | 8.23 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: TNF-alpha Levels in Patients Receiving Doxorubicin Containing Chemotherapy
Description: Continuous Measure of TNF-alpha at the 4 time points outlined in the protocol for each group.
Time Frame: prior to and 3 hours post doxorubicin and between cycles 1 and 2
Measure: Geometric Mean (95% Confidence Interval); unit: log(pg/ml)
Groups:
- Cycle 1 Saline; Cycle 2 Mesna: Saline infused over 15 minutes administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) during 1st cycle, then Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion during 2nd cycle
  Mesna: Mesna: 360 mg/m2 in 50 mL normal saline (NS) either on cycle 2 or cycle 1, day 1. Infused over 15 minutes
  Saline: Saline (used as a placebo) infused over the same time as mesna intervention
- Cycle 1 Mesna; Cycle 2 Saline: Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion during 1st cycle, then Saline administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) during 2nd cycle
  Mesna: Mesna: 360 mg/m2 in 50 mL normal saline (NS) either on cycle 2 or cycle 1, day 1. Infused over 15 minutes
  Saline: Saline (used as a placebo) infused over the same time as mesna intervention
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Number analyzed (Participants) | 16 | 16
log(pg/ml)
  Cycle 1 Pre | 3.55 [1.96 to 6.42] | 3.68 [1.98 to 6.81]
  Cycle 1 Post | 2.95 [1.54 to 5.64] | 3.18 [1.79 to 5.64]
  Cycle 2 Pre | 2.26 [1.37 to 3.73] | 1.67 [1.35 to 2.07]
  Cycle 2 Post | 1.78 [1.05 to 3.03] | 1.29 [1.01 to 1.65]
Statistical Analysis 1: Comparison: Cycle 1 Saline; Cycle 2 Mesna vs Cycle 1 Mesna; Cycle 2 Saline; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — This is for the interaction between baseline tnf-alpha levels and treatment received (mesna vs saline); Model was adjusted for baseline biochemical measures, time of measurement, treatment (mesna or saline), chemo type, and first-order interactions

2. Secondary Outcome: Protein Carbonyl Percent Changes From Baseline in Patients Receiving Doxorubicin Containing Chemotherapy
Description: Continuous Measure of percent changes from baseline of Protein Carbonyl at the 4 time points outlined in the protocol for each group. All measurements after naive baseline were adjusted as percent change from each individual's baseline measure.
Time Frame: prior to and 3 hours post doxorubicin and between cycles 1 and 2
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Number analyzed (Participants) | 16 | 16
Percent Change from Baseline
  Cycle 1 Post | 108.82 [88.20 to 134.26] | 73.54 [48.09 to 112.42]
  Cycle 2 Pre | 100.52 [79.52 to 127.07] | 97.00 [79.32 to 118.61]
  Cycle 2 Post | 87.91 [62.70 to 96.99] | 75.71 [49.81 to 115.08]

3. Secondary Outcome: Plasma HNE Percent Changes From Baseline in Patients Receiving Doxorubicin Containing Chemotherapy
Description: Continuous Measure of the percent change from baseline of Plasma HNE at the 4 time points outlined in the protocol for each group. All measurements after naive baseline were adjusted as percent change from each individual's baseline measure.
Time Frame: prior to and 3 hours post doxorubicin and between cycles 1 and 2
Measure: Geometric Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Number analyzed (Participants) | 16 | 16
Percent Change from Baseline
  Cycle 1 Post | 98.95 [89.06 to 109.94] | 102.63 [94.74 to 111.17]
  Cycle 2 Pre | 100.52 [79.52 to 127.07] | 97.00 [79.32 to 118.61]
  Cycle 2 Post | 87.91 [62.70 to 123.26] | 75.71 [49.81 to 115.08]

4. Secondary Outcome: Troponin Levels in Patients Receiving Doxorubicin Containing Chemotherapy
Description: Continuous Measure of troponin at the 4 time points outlined in the protocol for each group.
Time Frame: prior to and 3 hours post doxorubicin and between cycles 1 and 2
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Number analyzed (Participants) | 16 | 16
ng/ml
  Cycle 1 Pre | 0.015 [0.011 to 0.021] | 0.017 [0.013 to 0.021]
  Cycle 1 Post | 0.014 [0.010 to 0.019] | 0.012 [0.010 to 0.015]
  Cycle 2 Pre | 0.020 [0.014 to 0.029] | 0.016 [0.012 to 0.021]
  Cycle 2 Post | 0.021 [0.014 to 0.030] | 0.019 [0.014 to 0.026]

5. Secondary Outcome: B-type Natriuretic Peptide (BNP) Blood Levels in Patients Receiving Doxorubicin Containing Chemotherapy
Description: Continuous Measure of BNP at the 4 time points outlined in protocol for each of the groups. This is a 32-amino acid polypeptide secreted by heart ventricles in response to excessive stretching of cardiomyocytes.
Time Frame: prior to and 3 hours post doxorubicin and between cycles 1 and 2
Measure: Geometric Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Cycle 1 Saline; Cycle 2 Mesna | Cycle 1 Mesna; Cycle 2 Saline
Number analyzed (Participants) | 16 | 16
pg/ml
  Cycle 1 Pre | 46.36 [32.23 to 66.69] | 49.24 [33.00 to 73.48]
  Cycle 1 Post | 50.73 [34.16 to 75.35] | 47.17 [31.30 to 71.07]
  Cycle 2 Pre | 45.85 [36.19 to 58.08] | 46.30 [31.15 to 68.82]
  Cycle 2 Post | 54.33 [41.72 to 70.73] | 46.66 [32.03 to 67.97]

ADVERSE EVENTS:
Time Frame: All participants were followed clinically during first 2 cycles of therapy, for up to 24 weeks, and adverse events were assessed and classified using the Common Terminology Criteria for Adverse Events version 4.
Groups:
- Mesna: Mesna administered (infused over 15 minutes, 360 mg/m2) prior to and 3 hours post doxorubicin infusion during cycle assigned by randomization
  Mesna: Mesna: 360 mg/m2 in 50 mL normal saline (NS) on cycle 2, day 1. Infused over 15 minutes
- Saline: Saline administered prior to and 3 hours post doxorubicin infusion (over 15 minutes) during cycle assigned by randomization
  Infused over 15 minutes
Arm/Group | Mesna | Saline
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/32
Other Adverse Events (participants affected / at risk) | 29/32 | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesna (N=32) | Saline (N=32)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
MRSA positive infection in toe (Infections and infestations) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesna (N=32) | Saline (N=32)
Alanine aminotransferase increased (Investigations) | 4 (4) | 3 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9) | 15 (15)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Creatinine increased (Investigations) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Edema Limbs (General disorders) | 1 (1) | 2 (2)
Esophageal Spasms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (8) | 9 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoatremia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Lip Infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 10 (10) | 10 (10)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 12 (12) | 13 (13)
Neutrophil count decreased (Investigations) | 10 (10) | 9 (9)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 5 (5) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal Infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Weight Loss (Investigations) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 16 (16) | 9 (9)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
We did not measure any cognitive outcomes. We did not measure levels of anti-inflammatory cytokines, which could play a role in pathophysiology of Chemotherapy induced cognitive impairment (CICI). Small sample size, needs future trials to confirm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No